CLINICAL TRIAL: NCT01275820
Title: A Study to Evaluate Glucose and Insulin Response to Nutralin
Status: Completed | Type: Observational
Sponsor: Avera McKennan Hospital & University Health Center (Other)
Collaborators: Vintek, LLC (Unknown)
Responsible Party: Dave Kuper, RPh, Avera Research Institute
Other Study IDs: ARI-1330-Nutralin
Record Dates: First submitted 2011-01-10; First posted 2011-01-12 (Estimated); Last update posted 2011-01-12 (Estimated); Status verified 2011-01

CONDITIONS: Diabetes
Keywords: diabetes, insulin, blood sugar
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Nutralin: All 10 subjects in the study will consume the investigational food product.
  Interventions: Dietary Supplement: Nutralin

INTERVENTIONS:
Dietary Supplement: Nutralin — Food product to be taken 15 minutes prior to each of the three main meals of the day.
  Other Names: No other names at this time.

SUMMARY:
The purpose of this study is to evaluate how an investigational food product affects a healthy person's blood sugar and insulin levels.

DETAILED DESCRIPTION:
The investigational food product has helped decrease the amount of insulin needed in treating diabetic dogs and has improved the dogs' longevity and quality of life. Observational analysis by trained veterinarians has indicated that the natural fluctuations in blood glucose levels do not exist in dogs using the product. The hypothesis for this study is that healthy human subjects will have an increase in insulin levels after consuming the investigational food product.

ELIGIBILITY:
Inclusion Criteria:

* Men and women who are at least 18 years of age
* Non-diabetic

Exclusion Criteria:

* Diabetes
* Women who are pregnant, breastfeeding or planning to become pregnant
* Current and active liver or kidney disease
* Any food allergies
* Celiac disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals in and around the area of Sioux Falls, SD
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2010-06; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Glucose blood level | 4 weeks
  Measure the change in blood sugar levels

SECONDARY OUTCOMES:
Dosage of Insulin | 4 weeks
  Measure the levels of insulin

CONTACTS AND LOCATIONS:
Overall Officials: Edward Zawada, MD, Principal Investigator — Avera McKennan Hospital & University Health Center
Locations (1):
- Avera Research Institute, Sioux Falls, South Dakota, United States